CLINICAL TRIAL: NCT07019974
Title: Imposter Syndrome In Medical Students And Its Relationship With Stress
Brief Title: Imposter Syndrome in Medical Students and Its Relation With Stress
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Nimra Faraz, Dr, Rawalpindi Medical College
Other Study IDs: PH46 46 24
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Imposter Syndrome; Medical Students
MeSH Terms: conditions — imposter syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine the relationship between Imposter Syndrome and stress in undergraduate medical students at Rawalpindi Medical University, with particular attention to variables such as gender, academic year, and academic performance.

The main questions it aims to answer are:

Is there a positive correlation between Imposter Syndrome and stress?

Are gender and year of study associated with differences in stress and Imposter Syndrome levels?

Participants will:

Complete an online questionnaire including demographic questions

Fill out the Clance Impostor Phenomenon Scale (CIPS) to assess Imposter Syndrome

Complete the Perceived Stress Scale (PSS) to measure stress levels

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate MBBS students enrolled at Rawalpindi Medical University
* Students from any year of study (1st to final year)
* Willingness to participate, demonstrated by providing informed consent
* Ability to complete the online questionnaire independently

Exclusion Criteria:

* Postgraduate medical students or students from other disciplines (e.g., nursing, dentistry)
* Participants with known psychiatric diagnoses (e.g., depression, anxiety disorders) that could confound stress or Imposter Syndrome assessments
* Incomplete or partially filled questionnaires
* Students who did not consent to participate in the study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Undergraduate MBBS students enrolled at Rawalpindi Medical University
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Level of Imposter Syndrome among undergraduate medical students | May - August 2024
  The degree of Imposter Syndrome will be measured using the Clance Impostor Phenomenon Scale (CIPS). Participants will receive a total score based on their responses, which will be categorized as few characteristics, moderate, frequent, or intense. The outcome will help identify the prevalence and severity of Imposter Syndrome in the study population and will be analyzed in relation to stress, gender, and academic year.

CONTACTS AND LOCATIONS:
Overall Officials: Sumia Fatima, Dr, Study Chair — Rawalpindi Medical College
Locations (1):
- Rawalpindi Medical University, Rawalpindi, Punjab Province, Pakistan